CLINICAL TRIAL: NCT04473378
Title: Pilot Study of Glucose Monitoring to Determine Rates of Hyperglycemia During Chemotherapy for Early Stage Breast Cancer
Brief Title: Glucose Monitoring During Chemotherapy
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Melissa K Accordino, Assistant professor of medicine at CUMC, Columbia University
Other Study IDs: AAAS3402
Record Dates: First submitted 2020-07-13; First posted 2020-07-16 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer; Hyperglycemia
Keywords: Freestyle Libre Pro
MeSH Terms: conditions — Breast Neoplasms; Hyperglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- FreeStyle Libre sensor cohort: Patients with early stage breast cancer will have their blood glucose levels monitored by the Freestyle libre pro sensor.
  Interventions: Device: FreeStyle Libre Pro

INTERVENTIONS:
Device: FreeStyle Libre Pro — The device uses patches that attach to the skin on the back of the arm to measure blood sugar changes for the duration of the chemotherapy course.

SUMMARY:
This is a research study to look at blood sugar changes during chemotherapy using a continuous blood sugar monitoring device. The device uses patches that attach to the skin on the back of the arm to measure blood sugar changes for the duration of the chemotherapy course. Each patch lasts for about 2-weeks. During chemotherapy visits, new patches will be placed and will be worn until the chemotherapy course is complete. Participants will be in this study for 6 months. Approximately 50 patients will be enrolled in this study.

DETAILED DESCRIPTION:
This is a prospective observational cohort study monitoring trends in glucose in patients with early stage breast cancer treated with neoadjuvant or adjuvant chemotherapy. Patients will wear a noninvasive glucose monitoring sensor, the Freestyle Libre Pro for the duration of chemotherapy. The primary goal of this trial is to evaluate the prevalence of hyperglycemia in patients with early-stage breast cancer during neoadjuvant/adjuvant chemotherapy. Fifty patients will be enrolled. During each chemotherapy encounter, subjects will have their glucose sensor scanned in order to download subjects' glucose data. If the sensor has become no longer adherent to the participant's skin, participants will bring the sensor with them to the chemotherapy infusion center to be scanned. During each chemotherapy encounter, the Free Style Libre sensor will be replaced by the study team. Participants who receive chemotherapy every three weeks will be asked to come in 10-14 days after their chemotherapy infusion to replace the sensor. The sensors will be worn through completion of chemotherapy (the duration will vary based on the individual's chemotherapy regimen). Patients will have fructosamine, a glucose biomarker, and serum creatinine testing at baseline and every 3 weeks (weeks 3, 6, 9, 12, 15, 18, 21, 24) until week 24 (note: week 15, 18, and 21 are optional). Patients will have additional glucose biomarker testing (hemoglobin a1c, glucose, and insulin [fasting preferred]) at baseline, week 12 and week 24. Patients will also complete questionnaires assessing for symptoms of chemotherapy induced peripheral neuropathy, quality of life, and fatigue at baseline, week 12 and week 24. Visits will be conducted within the below specified windows forbidding unexpected circumstances such as missed appointments or loss to follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* History of stage I-III breast cancer
* Patient scheduled to receive adjuvant or neoadjuvant chemotherapy
* Signed informed consent

Exclusion Criteria:

* Current treatment with insulin
* Current treatment with non-topical steroids, with the exception of steroid treatment as a supportive chemotherapy medication
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with early stage breast cancer.
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2019-10-31 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-17 (Actual)

PRIMARY OUTCOMES:
Prevalence of hyperglycemia | 24 weeks
  assess the prevalence of HG, defined as the number of participants who have ≥1 glucose value of ≥140 mg/dL at any point during chemotherapy

SECONDARY OUTCOMES:
Prevalence of impaired glucose tolerance at baseline in nondiabetic patients. | Baseline
  Prevalence of glucose intolerance will be defined as a hemoglobin a1c >5.7% at baseline in nondiabetic patients The American Diabetes Association classifies individuals with a hemoglobin A1c level of 5.7-6.4% as having an increased risk of DM.The American Diabetes Association classified individuals with a hemoglobin A1c level of 6.5% or higher on two separate occasions as having a diagnosis of DM.
Patient-Reported Outcomes Measurement Information System (PROMIS)-29 | Baseline, week 12, and week 24
  The PROMIS-29 consists of 29 questions to measure global quality of life, including four questions from each of the following domains: anxiety, depression, fatigue, pain interference, physical function, sleep disturbance, satisfaction with participation in social roles, ability to participate in social roles and activities; it includes a single pain intensity item.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Accordino, MD, Principal Investigator — Columbia University
Locations (1):
- Herbert Irving Pavilion, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ulene SR, Wang S, Cook JR, McAuley F, Wooster ME, Faheem KF, Varoli A, McGuinness JE, Vasan N, Trivedi MS, Crew KD, Harden E, Law C, Hershman DL, Accordino MK. Continuous glucose monitoring to characterize hyperglycemia during chemotherapy for early stage breast cancer. Breast Cancer Res Treat. 2025 Aug;212(3):511-519. doi: 10.1007/s10549-025-07745-z. Epub 2025 Jun 4. PMID 40468140